CLINICAL TRIAL: NCT02614430
Title: Recover Working Life - Back on the Job After Acute Illness. A Study of the Effect on Functional Capacity and Self-rated Health and Working Capacity of a Vocational Training Course After Discharge From an Acute Hospitalisation
Brief Title: Recover Working Life - Back on the Job After Acute Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Amager Hospital (Other)
Responsible Party: Principal Investigator, Ove Andersen, Research Director, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GA-2015
Record Dates: First submitted 2015-10-09; First posted 2015-11-25 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Specific Work Inhibition
Keywords: Rehabilitation; Prediction; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vocational training (Active Comparator): Participants are randomized into the intervention group (training) where they are offered a training course of 4-9 weeks of physical training three times a week with a physiotherapist.
  Interventions: Other: Vocational training
- Control (No Intervention): Participants are randomized into the control group where they are offered the standard treatment.

INTERVENTIONS:
Other: Vocational training — The intervention consists of a physical training program, individual motivational talks and guidance on labor market-oriented topics. Each program is customised to the patient's physical resources and conditions where. The framework for the intervention of physical activity 1 hours 3 times weekly with concurrent motivational talks for an overall maximum duration of 9 weeks. Based on an assessment of the patient is instructed about pain management, ergonomics, conflict management, diet, lifestyle, behavior modification, stress symptoms and preventive home training.
  Arms: Vocational training

SUMMARY:
The project will investigate levels of physical, psychosocial functions and inflammatory biomarkers in a group of patients who by self-assessment indicates a perceived risk of decline in work ability after hospital admittance. The patients will be randomised to an intervention of physical training and followed for development in functional levels compared with patients not receiving the intervention. The goal is to validate measures of work ability assessment in connection to hospital admittance. The validation will provide important information about the quality of rehabilitation services that many municipalities provides through private suppliers - and where the effect on work ability lacks evidence-based documentation.

The project aims to link patient treatment to recovery and an optimal return to everyday life, comprising the patients work life. The frame is a multi-sectoral accepted platform for assessing patients' needs for care, treatment and rehabilitation, which is based on a professional assessment of the efficacy and quality of, varies heath care related deliveries. The acceptance of a multi-sectoral creates a need for accessible clinical tests of physical and mental functioning, combined with biomarkers to identify patients need.

The project investigates whether it is possible to identify patients (age 18 to 60 year) with an increased risk of losing their ability to work after discharge from an acute hospitalisation. And to evaluate whether measurable effects on inflammation and functional levels of labour oriented training program can be identified.

DETAILED DESCRIPTION:
The project will examine the validity of identification of patients in risk of decreased work ability during and after hospitalisation and the effect of early intervention on the physical and mental functional level. The project consists of a pilot study and two clinical studies investigating the following:

* The validity of work ability assessments by a self-administered questionnaire during hospitalisation.
* The development in the inflammatory response after discharge in relation to the development in self-rated health.
* The effect of a labour oriented training program measured in inflammatory response and functional level.
* The effect of a labour oriented training program on work ability after discharge.

The self-administered questionnaire Work Ability Index will be tested and evaluated during the pilot study.

Study 1 is a prospective cohort study testing the identification tool for decreased work ability including inflammatory biomarkers and functional levels after discharge.

Study 2 is a randomised controlled intervention study of the effect of a labour oriented training program initiated within 2 weeks after discharge on functional level and self-rated health.

Primary aim of study 1: testing the validity of Work Ability Index in relation to observations on functional level and measurement of inflammatory biomarkers after discharge.

Primary aim of study 2: examine the effect of labour oriented training on functional level and work ability.

Following measuring tools will be used during the project: Work Ability Index, hand grip strength, gait speed (6M), Major Depression Inventory (MDI), Self-rated health (EQ-5D) and inflammatory biomarkers including markers for inflammatory receptors, cytokines and chemokines.

Hand grip strength:

The project manager and trained clinical staff will test participants included in study 1. Participants are tested for physical capacity measured by grip strength. This is assessed twice by a hand dynamometer for 5 seconds with his dominant hand and an average is calculated.

Gait speed (6M):

Physical function is measured by a walking test of 6 m. The participants are measured from a starting line with the message to go in for them normal pace on a marked field of 8 m. The time is measured when the first foot reaches the 6m point and the test is repeated, after which an average is calculated.

Major Depression Inventory (MDI):

MDI is a depression questionnaire to 10 symptoms, which is part of the World Health Organization's definition of depression. The table focuses on the patient's current experience of symptoms within the last two weeks and the changes that the disease extent and rehabilitation can cause. MDI is used in the study as a rating scale with a theoretical sum score from 0 (no depression) to 50 (maximum depression).

EQ-5D:

EQ-5D is a validated questionnaire to measure health status by a simple descriptive profile and a single index value, which is evaluated for clinical and health economic studies of self-rated health. The questionnaire was approved by the EuroQol Group, and includes questions about mobility, personal care, activity, depression and pain.

Biomarkers:

At admission, 2 - and 12 weeks after discharge blood sample is taken for analysis of inflammatory receptors, cytokines and chemokines. The analyses will be carried out as batch after sample collection by ELISA and / or Luminex technology.

Total duration of the test, instruction and replies to the questionnaires represent a total of 45 minutes per. participant Patients who submit a written informed consent to participate based on an interview are randomised into an intervention or control group. The groups are stratified for hospitalisation due to medical and surgical reasons, physical work load and education to ensure an equitable distribution among participant receiving the intervention.

The intervention is performed in public-private collaboration with a health care provider specialised in labour oriented training. The program consists of a physical training program, individual motivational talks and guidance on labour market-oriented topics. Each program is customised to the patient's physical resources and conditions. The scope of the intervention is physical activity 1-2 hours 3 times weekly with concurrent motivational talks for an overall of max. 9 weeks.

The project aims to include 120 patients giving an interventions size of 50 participants and an estimated drop-out rate of 20%. The studies are carried out in accordance with the principles of the Helsinki Declaration.

Participants are covered by Amager Hvidovre Hospital Patient Insurance. The collected data will be kept in accordance to the Data Protection Agency guidelines.

The Project Manager will work with the clinical staff from the participating departments responsible for contacts with all patients who meet the inclusion criteria for the studies. Patients who meet the inclusion criteria will receive written and verbal information about the project including the advantages, disadvantages, risks and patient rights by participation in the project. The patient contacted by the project manager the day after the verbal and written information. If the patient wishes to participate in the project obtained accepted consent form and schedule time for tests and blood sampling.

Results:

The project will help to focus attention on an overlooked task in health care, where the patient after treatment can still be at risk of losing their ability to work. The project will also mean greater knowledge about the use of biomarkers and how these may reflect the development of the individual's refund and the current level of functioning.

ELIGIBILITY:
Inclusion Criteria:

* Acute medical/surgical patients between 18 to 60 years
* Patients who have been hospitalised for at least 12 hours
* Are entitled to sickness or unemployment benefits either from the employer or municipality
* Patients who have an increased risk of loss of earning capacity of> 50% relative for the total group of patients in the pilot study

Exclusion Criteria:

* Patients unable to cooperate
* Patients with end-stage disease
* Patients with major trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Day of recovery after sick leave | From discharge to 52 weeks after discharge
  Time to recovery date from discharge is defined the first day back at work after sick leave. Data on day of recovery will be subtracted from register kept by Statistics Denmark.

SECONDARY OUTCOMES:
Day of recovery after sick leave | From discharge to 12 weeks after discharge
  Time to recovery date from discharge is defined the first day back at work after sick leave. Data on day of recovery will be subtracted from register kept by Statistics Denmark.
Diagnose | From admission (Baseline) to 12 weeks after discharge
  Data on patient's diagnosis will be subtracted from the National Patients Registry in relation to ICD-10. This will be used to measure severity of disease.
SuPAR | From 2 weeks after discharge to 12 weeks after discharge
  Soluble urokinase plasminogen activator receptor: Biomarker of low-grade inflammation. SuPAR are measured 2 weeks- and 12 weeks after discharge.
Hand-grip strength of dominant hand | Admission (Baseline), 2 weeks after discharge and 12 weeks after discharge
  Development in isometric handgrip strength from 2 weeks to 12 weeks will be measured in the dominant hand using a handheld dynamometer (Digi-II; Saehan). The patient will be placed in a sitting position in an armchair, with the lower arm placed on the arm rest and an elbow flexion of 90 degrees. The patients will be asked to squeeze the handle as forcefully as possible for 5 secs. Handgrip strength will be expressed in kilograms.
Habitual gait speed | Admission (Baseline), 2 weeks after discharge and 12 weeks after discharge
  Development in physical function from 2 weeks to 12 weeks is measured by a walking test of 6 m. The participants are measured from a starting line with the message to go in for them normal pace on a marked field of 8 m. The time is measured when the first foot reaches the 6m point and the test is repeated, after which an average is calculated.
Major Depression Inventory (MDI) | Admission (Baseline), 2 weeks after discharge and 12 weeks after discharge
  MDI is a depression questionnaire to 10 symptoms, which is part of the World Health Organization's definition of depression. The table focuses on the patient's current experience of symptoms within the last two weeks and the changes that the disease extent and rehabilitation can cause. MDI is used in the study as a rating scale with a theoretical sum score from 0 (no depression) to 50 (maximum depression).
Health Related Quality of Life (EQ-5D) | Admission (Baseline), 2 weeks after discharge and 12 weeks after discharge
  EQ-5D is a validated questionnaire to measure health status by a simple descriptive profile and a single index value, which is evaluated for clinical and health economic studies of self-rated health. The questionnaire was approved by the EuroQol Group, and includes questions about mobility, personal care, activity, depression and pain. Low health-related quality is defined as below 80 on a scale of 0-100.
Work Ability Index (WAI) | From Admission (baseline), 2 weeks -, 12 weeks - and 52 weeks after discharge.
  Participants are tested for working capacity by answering WAI questionnaire, which in addition to self-assessed work contains parameters regarding self-rated health, marital status, education, smoking, alcohol and exercise.
  Low working capacity will be defined as patients who has; 1) a disease that affects the work capacity, 2) One or more doctor diagnosed diseases or 3) pain in muscles and joints.
Readmission | From discharge to 52 weeks after discharge
  Readmission is measured from the day of discharge to the day the patient is readmitted to a hospital. Data from the National Patients Register kept by the statistics Denmark will be subtracted.
Medication | From discharge to 12 weeks after discharge
  Data on medication use will be subtracted from National Prescription registry kept by Statistics Denmark. This will be used as an explanatory of a possible lack of effect on the primary outcome.
Doctor visits | From discharge to 52 weeks after discharge
  Data on visits to the doctor will be subtracted from register of National Health Insurance kept by Statistics Denmark. This will be used as an explanatory of a possible lack of effect on the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, PHD, MD, Principal Investigator — Clinical Research Centre, University Hospital of Copenhagen, Hvidovre
Locations (1):
- Clinical research Centre, Amager Hvidovre hospital, Hvidovre, Denmark